CLINICAL TRIAL: NCT02758327
Title: Evaluation of Tear Osmolarity Over Time With Sustained Use of Thera Tears Lubricating
Brief Title: Evaluation of Tear Osmolarity Over Time With Sustained Use of Thera Tears Lubricating Drops
Acronym: AKORN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Koffler Vision Group (Other)
Collaborators: Akorn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH_PM_101_14
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dry Eye Syndrome
Keywords: Tear Osmolarity; Keratitis Sicca; Ocular Surface Disease; TheraTears
MeSH Terms: conditions — Dry Eye Syndromes; Keratitis sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TheraTears Lubrication Drop (Experimental): TheraTears Lubricating Eye Drops to be instilled 1 drop in both eyes 4 times per day over a period of 8 weeks.
  Interventions: Drug: TheraTears Lubricating Eye Drops

INTERVENTIONS:
Drug: TheraTears Lubricating Eye Drops — Sodium Carboxy-methylcellulose 0.25% eye Lubricant
  Other Names: 87049747

SUMMARY:
The objective of the study is to demonstrate a change in osmolarity over time when moderate to severe dry eye subjects are treated with TheraTears lubricating drops.

DETAILED DESCRIPTION:
Symptomatic dry eye subjects exhibited a significantly higher tear osmolarity than observed in normal subjects, this is thought to relate to the inherent tear film instability of dry eye disease. Lubricating eye drops are frequently prescribed to relieve the symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 21 years of age and has full legal capacity to volunteer;
2. Has read and signed the information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is diagnosed with dry eye syndrome (in at least one eye), indicated by current ocular examination, prior history (self-reported history of dry eye is acceptable) and current use of treatments for dry eye;
5. Has a minimum osmolarity reading of 316 mosm/kg at the baseline visit in at least one eye or a osmolarity reading of at least 308 (in worse eye) and at least an 8 point difference between the two eyes.

Exclusion Criteria:

1. Has taken part in another research study within the last 30 days;
2. Planned contact lens wear during the course of the study;
3. Staff at the investigational site or family member of site staff or family member of currently enrolled participant;
4. Any subject that violates the washout period by using eye drops during the 72hrs washout period;
5. Has any known ocular disease* including active ocular infection, inflammation or allergy, especially Salzmann's nodular degeneration, symptomatic conjunctivochalasis, and fixation disparity syndrome;
6. Restasis use can be included if they have been on it for at least 3 months and are stable.Used Restasis (or similar topical medication) within the last 6 months;
7. Has a systemic condition that in the opinion of the investigator may affect the dry eye status of the subject, especially those newly diagnosed, newly prescribed and/or unstable;
8. Is pregnant, lactating or planning a pregnancy at the time of enrolment (verbal confirmation necessary);
9. Use of systemic anti-histamines, as long as they have been on them continuously for at least 1 month. Use of medications such as: Systemic Antihistamine (e.g., Allegra®, Benadryl®, Claritin®, Dimetapp®, Unisom®, Zyrtec®, etc.), Isotretinoin (e.g., Accutane®, Roaccutane®, Amnesteem®, Claravis®, Isotroin®, Sotret®) or similar medications;
10. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
11. Has undergone ocular surgery(LASIK, Cataract, etc)within the last year;

    * For purposes of this study, ocular conditions that are typically associated with dry eye status, such as meibomian gland dysfunction, mild (i.e. not considered clinically relevant) blepharitis, corneal and conjunctival staining are not considered an exclusion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Tear Osmolarity | 8 weeks
  Osmolarity measures will be evaluated using the eye with the highest osmolarity reading at the washout/baseline visit. These baseline values will be compared to subsequent follow-up visits, to determine change from baseline at each visit as well as cumulative change in osmolarity over time.

SECONDARY OUTCOMES:
Change in Visual Acuity | 8 weeks
  Visual acuity measures will be evaluated using the eye with the highest osmolarity reading at the washout/baseline visit. These baseline values will be compared to subsequent follow-up visits, to determine change from baseline at each visit as well as cumulative change in visual acuity over time.
Change in Tear Film Breakup Time | 8 Weeks
  After instillation of fluorescein, the investigator will ask the participant blink three times and keep their eyes open for as long as they can while the investigator records the time at which the dark spots on the tear film begin to appear.
Change in Corneal Staining | 8 weeks
  A fluorescein strip will be wetted with a few drops of saline, and applied to the inferior palpebral conjunctiva of both eyes. The eye will be illuminated by cobalt blue light, and viewed through a Wratten no. 12 barrier filter. Fluorescein staining will be assessed using the CCLRU8 scale (0 to 4).
Change in Conjunctiva Staining | 8 Weeks
  A lissamine green strip will be wetted and applied to the inferior palpebral conjunctiva of both eyes to assess conjunctival staining. Lissamine conjunctival staining will be assessed using the Oxford scale. If lissamine strip is not available, fluorescein maybe used instead to assess all conjunctival staining.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Houtman, MD, Study Director — Akorn Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided